CLINICAL TRIAL: NCT00266708
Title: Randomized Trial of Risedronate to Prevent Bone Loss in Renal Transplant
Brief Title: Randomized Trial of Risedronate to Prevent Bone Loss in Renal Transplant Recipients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-08-224
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Renal Transplant Osteodystrophy
Keywords: renal transplant; post-transplant osteoporosis
MeSH Terms: interventions — Risedronic Acid; Diphosphonates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Risedronate (Experimental): subjects received Risedronate for one year
  Interventions: Drug: Risedronate
- subjects received placebo (Placebo Comparator): subjects received placebo for 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risedronate — risedronate 35 mg weekly
  Other Names: bisphosphonate
  Arms: Risedronate
Drug: Placebo — Risedronate Placebo 35 mg weekly
  Other Names: Risedronate placebo
  Arms: subjects received placebo

SUMMARY:
Patients with kidney failure have underlying bone disease at the time of transplant. Fractures of various bones can be as high as 22%. Medication required for the transplant plays a role in bone loss.

Bisphosphonates are used in the general population to treat bone loss of osteoporosis and steroid-induced bone loss. While previous studies, using various bisphosphonates, have shown preservation of bone mineral density in renal transplant recipients, we have demonstrated that pamidronate, a second generation bisphosphonate, is associated with low bone turnover while still preserving bone mineral density. Improved bone mineral density is associated with decreased fracture risk in the general population, while low bone turnover may be associated with increased fracture in dialysis patients.

The purpose of this study is to determine whether risedronate, a third generation bisphosphonate, is effective in preserving bone density when given prophylactically following renal transplantation and whether it is associated with low bone turnover at one year following renal transplantation.

DETAILED DESCRIPTION:
Participants who receive a living donor kidney transplant undergo a bone biopsy at the time of kidney transplant and after one year of protocol. Once adequate kidney function is established, both groups take by mouth a weekly capsule (the control group has a placebo; the treatment group has risedronate 35 mg). Both groups undergo baseline, 6 month and 12 month dual energy x-ray absorptiometry (DEXA) bone mineral density scans. Both groups undergo bone hormonal studies at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adults with end stage renal disease who are undergoing living donor kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Coco, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Coco M, Pullman J, Cohen HW, Lee S, Shapiro C, Solorzano C, Greenstein S, Glicklich D. Effect of risedronate on bone in renal transplant recipients. J Am Soc Nephrol. 2012 Aug;23(8):1426-37. doi: 10.1681/ASN.2011060623. Epub 2012 Jul 12. PMID 22797188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Transplant candidates from Montefiore Medical Centre were recruited for the study.
Pre-assignment Details: 117 transplant candidates were identified as potentially eligible for the study. 57 of the 117 refused to participate and 60 of the candidates signed consent forms. Of the 60 who signed, 18 were either not transplanted or lost to follow-up so only 42 were randomized.
Groups:
- Risedronate: subjects received Risedronate for one year
  Risedronate 35 Mg: risedronate 35 mg weekly
- Placebo: subjects received placebo for 1 year
  Placebo weekly
Period: Overall Study
Arm/Group | Risedronate | Placebo
Started (Randomize) | 20 | 22
Completed | 16 | 13
Not Completed | 4 | 9
Not completed — No renal function | 1 | 1
Not completed — Refused biopsy | 3 | 6
Not completed — Asthma | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11) | 48 (14) | 44.7 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 16 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 3 | 6
  Hispanic | 10 | 11 | 21
  White | 5 | 6 | 11
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
BMD Calcium - Spine [Mean (Standard Deviation); unit: gm/cm^2] | 1.01 (0.17) | 1.01 (0.17) | 1.01 (0.17)
BMD Calcium - Hip [Mean (Standard Deviation); unit: gm/cm^2] | 0.90 (0.15) | 0.92 (0.17) | 0.909 (0.16)
BMD Calcium - Forearm [Mean (Standard Deviation); unit: gm/cm^2] | 0.54 (0.09) | 0.61 (0.09) | 0.57 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density of Spine at 6 Months
Description: Bone Mineral Density (BMD) measurements were of the vertebral spine (L1-L4) measured using the Hologic 4500 QDC scanner.
Time Frame: month 6 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 0.98 (0.16) | 0.97 (0.14)

2. Primary Outcome: Bone Mineral Density of Spine at 12 Months
Description: Bone Mineral Density (BMD) measurements were of the vertebral spine (L1-L4) measured using same Hologic 4500 QDC scanner.
Time Frame: month 12 of treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 1.00 (0.18) | 1.00 (0.18)

3. Primary Outcome: Bone Mineral Density of the Hip at 6 Months
Description: Bone mineral density (BMD) of the total hip were measured using the Hologic 4500 QDC scanner.
Time Frame: month 6 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 0.88 (0.13) | 0.86 (0.13)

4. Primary Outcome: Bone Mineral Density of the Hip at 12 Months
Description: Bone mineral density (BMD) of the total hip were measured using the Hologic 4500 QDC scanner.
Time Frame: month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 0.91 (0.13) | 0.87 (0.15)

5. Primary Outcome: Bone Mineral Density of Forearm at 6 Months
Description: Bone mineral density (BMD) of the distal third of the nondialysis access forearm were measured using the Hologic 4500 QDC scanner.
Time Frame: month 6 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 0.57 (0.11) | 0.58 (0.11)

6. Primary Outcome: Bone Mineral Density of Forearm at 12 Months
Description: as for outcome 5
Time Frame: month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: gm/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 20 | 22
gm/cm^2 | 0.55 (0.12) | 0.58 (0.09)

7. Secondary Outcome: Bone Histomorphometry - Percent Bone Volume (BV/TV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Percent Bone Volume is the percentage of total volume occupied by calcified bone. Percent Bone volume is calculated as Bone Volume (BV) divided by Tissue Volume (TV), where TV is bone plus marrow.
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 10.7 (6) | 13.3 (9)
  month 12 | 11.3 (5) | 9.7 (4)

8. Secondary Outcome: Bone Histomorphometry - Trabecular Thickness (TbTh)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. The ends of certain bones, known as cancellous bones, are actually not solid but are full of holes that are connected to each other by thin rods and plates of bone tissue known as trabeculae. Trabeculae of bone provide structural support to the spongy bone found at the ends of long bones. Trabeculae Trabecular Thickness (TbTh), a structural parameter, is the distance across individual trabecula.
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
micron
  Baseline | 72.6 (17) | 90.9 (39)
  month 12 | 72.1 (28) | 62.2 (20)

9. Secondary Outcome: Bone Histomorphometry - Percent Mineralized Bone Volume (MdV/BV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Percent Mineralized Bone Volume is the percentage of Bone Volume consisting of mineralized bone. Percent Mineralized Bone Volume is calculated as Mineralized Bone Volume (MdV) divided by Bone Volume (BV).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 95 (3) | 95 (4)
  month 12 | 92 (7) | 96 (6)

10. Secondary Outcome: Bone Histomorphometry - Mineralized Bone Volume (MdV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Bone mineralization is the process of laying down minerals on the matrix of the bone, with calcium and phosphorus as the most abundant minerals. Mineralized Bone Volume (MdV) is the percentage of mineralized bone tissue.
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 1.2 (0.4) | 1.3 (1)
  month 12 | 1.2 (0.5) | 1.0 (0.5)

11. Secondary Outcome: Bone Histomorphometry - Percent Osteoid Volume Relative to Bone Volume(OV/BV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoid is the unmineralized, organic portion of the bone matrix that forms prior to the maturation of bone tissue. The reported values indicates the percent of a given volume of bone that consists of unmineralized bone. It is equal to Osteoid Volume (OV) divided by Bone Volume (BV).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 4.1 (2.6) | 4.6 (3.4)
  month 12 | 8.7 (7.2) | 4.9 (5)

12. Secondary Outcome: Bone Histomorphometry - Percent Osteoid Volume Relative to Tissue Volume (OV/TV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoid is the unmineralized, organic portion of the bone matrix that forms prior to the maturation of bone tissue. The reported values indicates the percent of a given volume of tissue (bone + marrow) that consists of unmineralized bone. It is equal to Osteoid Volume (OV) divided by Tissue Volume (TV).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 0.49 (0.4) | 0.58 (0.58)
  month 12 | 0.90 (0.8) | 0.51 (0.8)

13. Secondary Outcome: Bone Histomorphometry - Percent Osteoid Surface Relative to Bone Surface (OS/BS)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoid is the unmineralized, organic portion of the bone matrix that forms prior to the maturation of bone tissue. The reported values indicates the percent of bone surface that consists of unmineralized bone. It is equal to Osteoid Surface (OS) divided by Bone Surface (BS).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 23 (18) | 15 (8)
  month 12 | 24 (27) | 14 (10)

14. Secondary Outcome: Bone Histomorphometry - Percent Osteoblasts Relative to Bone Surface (OB/BS)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoblasts (OB) are cells that make bones by producing a matrix that becomes mineralized. Bone mass is a balance between the osteoblasts (OB) that form the bone and cells called osteoclasts (OC) that break down the bone. The reported values indicate the percent of bone surface (BS) that is made up of osteoblasts (OB).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 2.3 (3) | 1.3 (1.3)
  month 12 | 1.23 (1.6) | 0.75 (0.76)

15. Secondary Outcome: Bone Histomorphometry - Percent Osteoclasts Relative to Bone Surface (OC/BS)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoclasts (OC) are cells responsible for bone resorption, which is the breaking down of bones. Osteoclasts make and secrete digestive enzymes that break up or dissolve the bone tissue. Bone mass is a balance between the osteoblasts (OB) cells that form the bone and the osteoclasts (OC) cells that break down the bone. The reported values indicate the percent of bone surface (BS) that consists of osteoclasts (OC).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 16
percent
  Baseline | 1.5 (1.9) | 0.97 (1.2)
  month 12 | 0.28 (0.43) | 0.68 (1.23)

16. Secondary Outcome: Bone Histomorphometry - Percent Eroded Surface Relative to Bone Surface (ES/BS)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoclasts (OC) are cells responsible for bone resorption, which is the breaking down of bones. Osteoclasts make and secret digestive enzymes tha break up or dissolve the bone tissue. An eroded surface (ES) is the surface of the lacuna ( a cavity or depression in the bone) generated by an active OC. The reported values indicate the percent of eroded surface relative to bone surface (BS).
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
percent
  Baseline | 9 (11) | 1.36 (1.7)
  month 12 | 2.7 (3) | 0.82 (1.4)

17. Secondary Outcome: Bone Histomorphometry - Bone Formation Rate
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoblasts (OB) are cells that make bones by producing a matrix that becomes mineralized. Bone formation rate (BFR) indicates how much of the bone is actively mineralizing; it is determined by the number of active OB and the average work of each OB.
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: micron/day
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
micron/day
  Baseline | 0.02 (0.05) | 0.04 (0.1)
  month 12 | 0.10 (0.16) | 0.05 (0.06)

18. Secondary Outcome: Bone Histomorphometry - Osteoid Volume (OV)
Description: Bone histomorphometry is quantitative information on bone remodeling and structure, obtained through examination of an undecalcified bone biopsy. Osteoid is the unmineralized, organic portion of the bone matrix that forms prior to the maturation of bone tissue. The reported values indicates the Osteoid Volume (OV), the volume of bone that consists of unmineralized bone.
Time Frame: Baseline and month 12 of the treatment
Population: Calculation done on intent-to-treat population
Measure: Mean (Standard Deviation); unit: micron^3
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 16 | 13
micron^3
  Baseline | 0.06 (0.04) | 0.06 (0.06)
  month 12 | 0.10 (0.09) | 0.03 (0.02)

ADVERSE EVENTS:
Time Frame: Adverse events collected during course of study, which lasted 6 years.
Arm/Group | Risedronate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risedronate (N=20) | Placebo (N=20)
deep venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) — venous thrombosis and Blood clots that develop in a vein, usually in the leg or thing. It can cause pain and swelling in the leg and may lead to complications such as pulmonary embolism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes